CLINICAL TRIAL: NCT05716568
Title: Patient Tailored Contrast Volume for Preoperative CT Angiography of the Aorta: A Prospective Study Based on Patient Heart Rate and Body Surface Area Differences
Brief Title: Patient Tailored Contrast Volume for Preoperative CT Angiography of the Aorta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S58042
Record Dates: First submitted 2015-12-15; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2015-12

CONDITIONS: Aortic Aneurysm
Keywords: CT-angiography; Aortic aneurysm; Aortic dissection; Pre-operative; Contrast dose reduction
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard contrast dose (Active Comparator): Standard contrast dose administration
  Interventions: Other: Contrast dose reduction, CT-angiography
- Calculated contrast dose (Active Comparator): Contrast dose by calculation
  Interventions: Other: Contrast dose reduction, CT-angiography
- Calculated contrast dose -50% (Active Comparator): Contrast dose by calculation, with extra dilution by 50%.
  Interventions: Other: Contrast dose reduction, CT-angiography

INTERVENTIONS:
Other: Contrast dose reduction, CT-angiography — Contrast dose reduction for CT-angiography in pre-operative aorta

SUMMARY:
An in-house calculator was developed to calculate the appropriate contrast dose, rather than standardly administering a 120ml dose. This study aims for a more uniform contrast enhancement in patients by means of adjusting (lowering) contrast dose to patient parameters.

DETAILED DESCRIPTION:
Until now, CT scans in our and many other institutions are being performed with a fixed standard contrast dose specific for every protocol, independent of patient characteristics. However, many if not all patients would benefit from a contrast dose reduction, as long as image quality is not impaired. This is especially beneficial to patients with impaired renal function.

For this purpose, we researched previous literature as well as data from previously scanned patients with standard dose, to formulate a contrast dose calculation adapted to patient parameters.

An in-house calculator was developed to calculate the optimal contrast dose dependent on patient length, weight and heartrate.

A total of 60 CT-scans will be performed and retrospectively collected. Patients are randomly assigned to one of three groups : 1/ Standard dose of 120ml; 2/ Calculated dose (40-150ml) 3/ Calculated dose -50% (20-120ml). In case of reduced kidney function, patients were randomly divided between group 2 and 3 (reduced contrast dose).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring CT-angiography of the aorta as requested by clinician
* For aneurysm detection or follow-up
* Or for dissection follow-up
* Thoraco-abdominal aorta or abdominal aorta

Exclusion Criteria:

* Contra-indications for contrast administration (severe renal impairment or adverse reactions)
* Previously endovascular repair of the aorta
* Only thoracic aorta
* No informed consent
* Contrast injection at 4cc/second not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction in contrast dose | Through study completion, an average of 1 year
  Reduction in contrast dose while maintaining image quality

CONTACTS AND LOCATIONS:
Overall Officials: Geert Maleux, Prof Dr, Principal Investigator — Universitaire Ziekenhuizen KU Leuven